CLINICAL TRIAL: NCT03643991
Title: Decreasing Agitation in Patients With Dementia Through the Use of Weighted Blankets: A Pilot Study
Brief Title: Decreasing Agitation in Patients With Dementia Through the Use of Weighted Blankets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Maria I. Lapid, M.D., Principle Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-009951
Record Dates: First submitted 2018-08-20; First posted 2018-08-23 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Dementia
Keywords: Agitation; Dementia; Inpatient
MeSH Terms: conditions — Dementia; Psychomotor Agitation

STUDY DESIGN:
Intervention Model Description: Enrolled patients will be computer randomized in 1:1 ratio to either the intervention group or the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weighted Blanket Cohort (Experimental): Subjects will receive weighted blanket for three nights with monitoring by nurse. Weight of blanket is determined by weight of the patient (10% of patients body weight).
  Interventions: Other: Weighted Blanket
- Control Cohort (No Intervention): Subjects will receive treatment as usual while inpatient, no blanket.

INTERVENTIONS:
Other: Weighted Blanket — Weighted blanket will be given to patients based on the patient weight (10% of patients body weight) for three nights while on inpatient unit.
  Arms: Weighted Blanket Cohort

SUMMARY:
The purpose of this research study is to determine whether the use of weighted blankets help reduce behavioral and psychological symptoms, including agitation in people with dementia.

DETAILED DESCRIPTION:
The Intervention Group

1. Patient or Legally Authorized Representative (LAR) will be asked to sign a consent form and will have the study explained.
2. Nursing staff will complete baseline assessments to measure behavioral disturbances using the CMAI and CGI and other distressing symptoms using the ESAS-r.
3. A weighted blanket, based on admission body weight, will be provided to the patient under nursing supervision.
4. For 3 consecutive days after each use of weighted blanket, nursing staff will complete morning assessments to measure behavioral disturbances using the CMAI and CGI and other distressing symptoms using the ESAS-r.
5. At the end of the intervention, nursing staff will complete post-intervention assessments to measure behavioral disturbances using the CMAI and CGI and other distressing symptoms using the ESAS-r.

Control Group:

1. Patient or Legally Authorized Representative (LAR) will be asked to sign a consent form and will have the study explained.
2. The study team will recruit a group of patients with similar characteristics as described in the inclusion criteria; however, the patient will not receive the weighted blanket, but undergo the same assessments as described in 1-5 (above) and in the Schedule of Assessments.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted on the inpatient geriatric psychiatry unit, complex interventions unit, internal medicine service and/or admitted hospice GIP
* Documented diagnosis of dementia or suspected major neurocognitive disorder.
* Presence of agitation/aggression symptoms as defined by a minimum aggression score on the Cohen-Mansfield Agitation Inventory Short Version (CMAI): Patients must score 3, 4, or 5 on at least one question related to aggression (items 1-4).
* Have a LAR able to sign the consent on behalf of the patient.

Exclusion Criteria:

* Severe pain likely to be exacerbated by use of weighted blanket
* Inability to remove blanket;
* Skin burns or open wounds;
* Admitted on 72 hour hold.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Cohen-Mansfield Agitation Inventory Short Version (CMAI) Change | At baseline, days 1-3, and then within 72 hours of last use of the weighted blanket
  Assess the agitation/aggression outcome using numeric scales ranging from 1-5. The sum of the scores is defined as the agitation/aggression outcome and ranges from 14-70, with the lower score being the better outcome.

SECONDARY OUTCOMES:
The revised Edmonton Symptom Assessment System Revised (ESAS-r) Change | At baseline and within 72 hours of the last use of the weighted blanket.
  Assessment of symptoms in palliative patients using numeric analog scales ranging from 0 to 10 to assess levels of pain, tiredness, drowsiness, nausea, appetite, shortness of breath, depression, anxiety, and well-being. The sum of the scores for all symptoms is defined as the symptom distress score. The range of the sum is 0-100, with a lower score indicating a better outcome. The ESAS-r is a validated tool and publicly available for use.
Clinical Global Impressions (CGI) | At baseline, days 1-3, and then within 72 hours of last use of the weighted blanket
  Aggression/Agitation as a measure of the global clinical outcome using a numeric scale ranging from 1-7, with a lower score indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Lapid, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schenzel HA, Palmer AK, Shah NB, Lawson DK, Fischer KM, Lapid MI, DeFoster RE. Weighted Blankets for Agitation in Hospitalized Patients with Dementia: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Feb 26;14:e57264. doi: 10.2196/57264. PMID 40009836
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials